CLINICAL TRIAL: NCT07132723
Title: Associations Between Time to Reduction and Complications in Patients With Dislocated Total Hip Arthroplasty - A Protocol for an Observational Cohort Study
Brief Title: Associations Between Time to Reduction and Complications in Patients With Dislocated Total Hip Arthroplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HIP_REDUCTION
Record Dates: First submitted 2025-02-25; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-02

CONDITIONS: Closed Reduction; Arthroplasty, Replacement, Hip; Length of Stay
MeSH Terms: interventions — Time; Airway Management; Neuromuscular Blocking Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients underwent closed reduction of dislocated THA: adults presenting with a dislocated THA, who underwent closed reduction in an operating theatre with anesthesiology being involved, in public hospitals
  Interventions: Other: Time in minutes from admission to closed reduction

INTERVENTIONS:
Other: Time in minutes from admission to closed reduction — Time in minutes from admission to closed reduction measured as: From arriving time in the emergency department until the start of surgery in the operating theater.
  Other Names: - Time of day; - Weekday vs. weekend; - Airway management; - Anesthesia method(s); - Neuromuscular blocking agent (Yes/No)

SUMMARY:
The aim of the study is to investigate the impact of time to closed reduction on both patient related and organizational factors. These include, length of stay, hospitalization, admission to intensive care unit, rehospitalizations, delirium, all-cause mortality, infection requiring hospital contact, and cardiovascular complications. It is also intended to investigate whether different anaesthetic strategies and airway management are associated with different complication rates.

It is hypothesized that longer waiting time until reduction increase the postoperative length of stay, readmissions, and risk of complications.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered eligible for inclusion if they meet all of the following criteria:

* Aged 18 years or older
* Presented to the emergency department with a dislocated total hip arthroplasty.
* Undergo closed reduction of the dislocated total hip arthroplasty in the operating theatre, with the involvement of the Department of Anesthesiology.

Exclusion Criteria:

* Were primarily booked for open surgical reduction.
* Did not have a complete case log (i.e. time of admission; referral to the operation theatre; anesthesia induction; discharge, etc.) and we were unable to recreate the log using simple code rules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort contains all adults presenting with a dislocated THA, who underwent closed reduction in an operating theatre with anesthesiology being involved, in public hospitals in the Capital and Zealand Regions of Denmark.
  The study population is extracted from a dataset retrieved from the Electronic Health Record (EHR) system 'Sundhedsplatformen' (Epic Systems Corporation, WI, USA) from 1 January 2017 to 31 December 2024, including granular data from approximately 1.1 million anesthetic procedures
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Post procedure length of stay | 30 days after the closed reduction
  Post procedure length of stay from closed reduction until discharge from the hospital (hours)

SECONDARY OUTCOMES:
All-cause mortality | 90 days after closed reduction
  90 days all-cause mortality (Y/N)
Admissions to Intensive care unit | 30 days after the closed reduction
  Admissions to the intensive care unit within 30 days after the closed reduction.
Readmission | 30 days after discharge
  Readmission within 30 days after discharge
Delirium during admission | From admission to discharge up to 30 days after closed reduction
  Defined as diagnose of delirium (F05.x, obtained from the diagnosis codes from the given admission) or the non-planned administration of haloperidol, olanzapine, risperidone, or quetiapine (as a surrogate for new onset delirium)
Acute kidney failure | Post procedure until 30 days after discharge
  Defined as serum creatinine increase of more than 25 μmol/L within a period of less than 48 hours. (As a surrogate for acute kidney failure)
Infection requiring hospital contact | Post procedure until 30 days after discharge
  Defined as diagnosed infection (postoperative infection (T81.4), pneumonia (J13.x-J18.x), Cystitis (N30.x, N39.0), sepsis (R65.x A40.x, A41.x), C. difficile (A04.7) obtained from the diagnose codes from the given admission) or administration of antibiotic treatment (as a surrogate for in-hospital infection
Cardiovascular complications | From admission to 30 days after discharge.
  Defined as diagnosed arrythmia (I47.x, I48.x, I49.x), myocardial infarction (I21.x, I22.x), cerebral ischemia (I61.x, I63.x, I64.x), hemorrhage(T81), pulmonary embolism(I26.x) or deep venous thrombosis(I80.2) (obtained from the diagnosis codes from the given admission)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, North Zeeland Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT07132723/Prot_SAP_000.pdf